CLINICAL TRIAL: NCT02733627
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 1467335 in Healthy Male and Female Subjects (Double-blind, Randomised, Placebo-controlled Within Dose Groups)
Brief Title: To Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BI 1467335 Following Multiple Dose Administration Over 28 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1386.8; 2015-005049-29 (EudraCT Number)
Record Dates: First submitted 2016-03-30; First posted 2016-04-11 (Estimated); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- BI 1467335 10 mg (low dose) (Experimental)
  Interventions: Drug: BI 1467335
- BI 1467335 15 mg (medium dose) (Experimental)
  Interventions: Drug: BI 1467335
- BI 1467335 20 mg (high dose) (Experimental)
  Interventions: Drug: BI 1467335
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1467335
  Arms: BI 1467335 10 mg (low dose); BI 1467335 15 mg (medium dose); BI 1467335 20 mg (high dose)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 1467335 in healthy male and female subjects following oral administration of multiple rising doses over 28 days.

Secondary objectives are the exploration of the pharmacokinetics (PK) and target engagement biomarkers of BI 1467335 after multiple dosing.

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs, Blood pressure (BP), Pulse rate (PR), 12-lead Electrocardiogram (ECG), and clinical laboratory
* Age of 18 to 50 years (incl.)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects, or female subjects who meet any of the following criteria starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion:
* Surgically sterilised (including hysterectomy)
* Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of Follicle Stimulating Hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion criteria:

* Any finding in the medical examination (including Blood pressure(BP),Pulse rate (PR) or Electrocardiogram (ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication
* Used nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff) within 6 weeks before screening and unable to abstain from using these products until study completion
* Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/corrected QT (QTc) interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Detection of cataract in slit lamp examination
* GFR according to CKD-EPI-Formula < 90 mL/min at screening
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a double-blind, randomised, placebo-controlled within parallel dose groups, multiple dose trial.Only male subjects & postmenopausal or surgically sterilised female subjects were included into trial because at time of trial start-up no data on reproductive toxicology were available.
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated.
Groups:
- BI 1467335 10 mg (Low Dose): Participants were orally administered 20 ml solution containing 10 mg of BI 1467335: (0.5 mg/ml) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h).
- BI 1467335 15 mg (Medium Dose): Participants were orally administered 30 ml solution containing 15 mg of BI 1467335: (0.5 mg/ml) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h).
- BI 1467335 20 mg (High Dose); Placebo: Participants were orally administered 40 ml solution containing 20 mg of BI 1467335: (0.5 mg/ml) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h).
Period: Overall Study
Arm/Group | BI 1467335 10 mg (Low Dose) | BI 1467335 15 mg (Medium Dose) | BI 1467335 20 mg (High Dose) | Placebo
Started | 9 | 9 | 9 | 9
Completed | 9 | 8 | 7 | 9
Not Completed | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Withdrawn due laboratory reason concerning neutrophils in agreement with the sponsor | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All participants who received at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1467335 10 mg (Low Dose) | BI 1467335 15 mg (Medium Dose) | BI 1467335 20 mg (High Dose) | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: TS
  Years | 39.7 (7.9) | 33.8 (8.0) | 35.2 (8.4) | 38.7 (9.8) | 36.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: TS
  Participants
    Female | 3 | 1 | 1 | 3 | 8
    Male | 6 | 8 | 8 | 6 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: TS
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 9 | 9 | 9 | 9 | 36
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: TS
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 1 | 0 | 1
    White | 9 | 9 | 7 | 9 | 34
    More than one race | 0 | 0 | 1 | 0 | 1
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Investigator Defined Drug-related Adverse Events
Description: Number of subjects with investigator defined drug-related adverse events (AEs) is reported.
Time Frame: From first day of study drug administration until 20 days after last dose of study drug administration, up to 48 days.
Population: Treated set (TS): All participants who received at least 1 dose of trial medication.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 1467335 10 mg (Low Dose) | BI 1467335 15 mg (Medium Dose) | BI 1467335 20 mg (High Dose) | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 3 | 4 | 6 | 4

2. Secondary Outcome: Cmax
Description: Cmax is the maximum measured concentration of BI 1467335 in plasma after administration of the first dose.
Time Frame: 0:00 hour (h) (within 30 minutes prior to dosing) and 0:15 h, 0:30 h, 0:45 h, 1:00 h, 1:30 h, 2:00 h, 3:00 h, 4:00 h, 6:00 h, 8:00 h, 10:00 h, 12:00 h and 24:00 h after drug administration on Day 1.
Population: Pharmacokinetic parameter analysis set (PKS): All participants of the TS who provided at least 1 pharmacokinetic (PK) parameter that was not excluded due to relevant protocol violations or due to PK non-evaluability. Participants of the "Placebo" arm were not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/Liter (nmol/L)
Arm/Group | BI 1467335 10 mg (Low Dose) | BI 1467335 15 mg (Medium Dose) | BI 1467335 20 mg (High Dose)
Number analyzed (Participants) | 9 | 9 | 9
nanomol/Liter (nmol/L) | 1.79 (45.9) | 9.74 (30.6) | 25.0 (59.5)
Statistical Analysis 1: Comparison: BI 1467335 10 mg (Low Dose) vs BI 1467335 15 mg (Medium Dose) vs BI 1467335 20 mg (High Dose); The basic model for the investigation of dose proportionality was a power model. The model consisted of a regression model applied to log-transformed data. The corresponding ANCOVA model included the logarithm of the dose as a covariate. The assumption of a linear relationship between the log-transformed pharmacokinetic endpoint and the log-transformed dose was checked; Test type: Other; Slope = 3.8266, 95% CI 2-sided [3.2155 to 4.4376], Standard Error of Mean 0.2967; Standard Error of the mean is actually Standard Error of the slope. Based on the estimate for slope parameter (β), a 2-sided 95% CI for the slope was computed. Perfect dose proportionality would correspond to a slope of 1

3. Secondary Outcome: AUC0-24
Description: AUC0-24 is the area under the concentration-time curve of BI 1467335 in plasma over the time interval from 0 to 24 hours after administration of the first dose.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameter analysis set (PKS): All participants of the TS who provided at least 1 pharmacokinetic (PK) parameter that was not excluded due to relevant protocol violations or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol*hour/Liter (nmol*h/L)
Arm/Group | BI 1467335 10 mg (Low Dose) | BI 1467335 15 mg (Medium Dose) | BI 1467335 20 mg (High Dose)
Number analyzed (Participants) | 8 | 8 | 9
nanomol*hour/Liter (nmol*h/L) | 2.34 (61.2) | 17.0 (40.6) | 41.6 (39.7)
Statistical Analysis 1: Comparison: BI 1467335 10 mg (Low Dose) vs BI 1467335 15 mg (Medium Dose) vs BI 1467335 20 mg (High Dose); [analysis description as in outcome 2, analysis 1]; Test type: Other; Slope = 4.1810, 95% CI 2-sided [3.5094 to 4.8527], Standard Error of Mean 0.3247; [other analysis details as in outcome 2, analysis 1]

4. Secondary Outcome: Cmax,28
Description: Cmax,28 is the maximum measured concentration of BI 1467335 in plasma following administration of the 28th dose.
Time Frame: 648:00 hours (h) (within 30 minutes prior to dosing) and 648:15 h, 648:30 h, 648:45 h, 649:00h, 649:30 h, 650:00 h, 651:00 h, 652:00 h, 654:00 h, 656:00 h, 658:00 h, 660:00 h, 672:00 h after first drug administration on Day 1.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/Liter (nmol/L)
Arm/Group | BI 1467335 10 mg (Low Dose) | BI 1467335 15 mg (Medium Dose) | BI 1467335 20 mg (High Dose)
Number analyzed (Participants) | 9 | 8 | 7
nanomol/Liter (nmol/L) | 72.1 (71.0) | 189 (15.3) | 255 (24.6)
Statistical Analysis 1: Comparison: BI 1467335 10 mg (Low Dose) vs BI 1467335 15 mg (Medium Dose) vs BI 1467335 20 mg (High Dose); [analysis description as in outcome 2, analysis 1]; Test type: Other; Slope = 1.8868, 95% CI 2-sided [1.2503 to 2.5234], Standard Error of Mean 0.3069; [other analysis details as in outcome 2, analysis 1]

5. Secondary Outcome: AUC0-24,28
Description: AUC0-24,28 is the area under the concentration-time curve of BI 1467335 in plasma over the time interval from 0 to 24 hours after administration of the 28th dose.
Time Frame: 648:00 hours (h) (within 30 minutes prior to dosing) and 648:15 h, 648:30 h, 648:45 h, 649:00 h, 649:30 h, 650:00 h, 651:00 h, 652:00 h, 654:00 h, 656:00 h, 658:00 h, 660:00 h and 672:00 h after first drug administration on Day 1.
Population: Pharmacokinetic parameter analysis set (PKS): All participants of the TS who provided at least 1 pharmacokinetic (PK) parameter that was not excluded due to relevant protocol violations or due to PK non-evaluability. Participants of the "Placebo" arm were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol*hour/Liter (nmol*h/L)
Arm/Group | BI 1467335 10 mg (Low Dose) | BI 1467335 15 mg (Medium Dose) | BI 1467335 20 mg (High Dose)
Number analyzed (Participants) | 9 | 8 | 7
nanomol*hour/Liter (nmol*h/L) | 373 (143) | 1720 (12.8) | 2940 (29.5)
Statistical Analysis 1: Comparison: BI 1467335 10 mg (Low Dose) vs BI 1467335 15 mg (Medium Dose) vs BI 1467335 20 mg (High Dose); [analysis description as in outcome 2, analysis 1]; Test type: Other; Slope = 3.0677, 95% CI 2-sided [2.0631 to 4.0723], Standard Error of Mean 0.4844; [other analysis details as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: From first day of study drug administration until 20 days after last dose of study drug administration, up to 48 days.
Description: Treated set (TS): All participants who received at least 1 dose of trial medication.
Arm/Group | Placebo | BI 1467335 10 mg (Low Dose) | BI 1467335 15 mg (Medium Dose) | BI 1467335 20 mg (High Dose)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 7/9 | 4/9 | 8/9 | 7/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | BI 1467335 10 mg (Low Dose) (N=9) | BI 1467335 15 mg (Medium Dose) (N=9) | BI 1467335 20 mg (High Dose) (N=9)
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 0 | 2
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 3 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 3 | 3 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Apathy (Psychiatric disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT02733627/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT02733627/SAP_001.pdf